## SHORT TERM AND LONG TERM FOLLOW-UP RESULTS OF NEWBORNS WITH TRACHEOSTOMY

Document Date: June 10, 2020

## **Study Protocol (Follow-up Results of Newborns With Tracheostomy):**

In our study, the babies who were hospitalized in Hacettepe University İhsan Doğramacı Children's Hospital Department 37 Section 39 Neonatal Intensive Care Unit between 01.01.2005-01.06.2020, tracheostomy procedure and monitored at risky neonatal outpatient clinic will be scanned retrospectively by accessing their files from the computer database. The data will be added to the case report form.

## Inclusion Criteria:

These are the babies who stayed in Hacettepe University Ihsan Dogramaci Children's Hospital Neonatal Intensive Care Unit between 01.01.2005-31.12.2019, underwent tracheostomy procedure and followed up at risky neonatal outpatient clinic.

## **Exclusion Criteria:**

Newborns whose file and follow-up information required for the study are not available

We planned to determine the results of the study whether these babies should be careful in the follow-up and to take precautions in order to lead a better and healthier life, and what we can do in order to provide these babies and their families with better health care support.